CLINICAL TRIAL: NCT05823324
Title: The Effect of Therapeutic Play on Children's Pain, Anxiety, and Mothers' Anxiety During Peripheral Intravenous Catheterisation
Brief Title: The Effect of Therapeutic Play During Peripheral Intravenous Catheterisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Seda Caglar, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SeCaglar
Record Dates: First submitted 2023-03-28; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Pain; Anxiety
Keywords: pain; anxiety; Peripheral intravenous catheterisation; therapeutic play
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic play (Experimental): The therapeutic play method with the teddy bear during PIVC was applied in this group
  Interventions: Behavioral: Therapeutic play group
- Control (No Intervention): The standard procedure of the clinic was applied in the control group. The routine invasive procedure of the clinic, the mothers accompany their children and are involved in the procedure

INTERVENTIONS:
Behavioral: Therapeutic play group — The dramatization method with teddy bear, one of the TP methods, was applied during the PIVC intervention
  Arms: Therapeutic play

SUMMARY:
Therapeutic play (TP) is a non-pharmacological method used in the pain management in children. This study was conducted to determine the effect of therapeutic play on children's pain, anxiety, and mothers' anxiety during peripheral intravenous catheterisation (PIVC).

DETAILED DESCRIPTION:
The hospitalisation of children due to an acute or chronic illness interrupts play, disrupts their daily routines, places them in an unfamiliar environment, forces them to encounter with unfamiliar people, exposes them to invasive procedures, and makes them suffer from pain and anxiety. Peripheral intravenous catheterisation (PIVC) is probably the most common procedure performed in paediatric clinics. It has been estimated that 80% of hospitalised children have a peripheral intravenous catheter in place. PIVC is a painful and traumatic experience that children usually go through for the first time and frequently during the hospitalisation. This experience of children impairs effective communication between them and healthcare professionals and also causes problems in adaptation to the care and treatment process in the hospital setting. As one of the non-pharmacological pain relief methods, therapeutic play (TP) is a distraction that is defined as "the directed use of toys and materials, which can facilitate children to gain knowledge about the environment and the world they live in, to improve their perceptions thereof and to gain control, for a specific purpose". In order to call play with a child who is hospitalised as therapeutic, the play should encourage children to express their feelings and thoughts during the hospitalisation, assume an educational role in their positive or negative hospital experiences, and bring psychosocial and physical benefits. Children could be told facts such as the hospitalisation, the procedures to be followed and the time when this procedure would end through therapeutic play

ELIGIBILITY:
Inclusion Criteria:

* 3-6 year-old children,
* had no mental disability,
* were able to communicate,
* and had mothers volunteered to participate

Exclusion Criteria:

* none

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change from before in pain on the FLACC Scale at during peripheral intravenous catheterisation | data collected just before and within 5 min after peripheral intravenous catheterization procedure
  The FLACC Scale was used to assess the pain scores of children. The scale is scored between 0 and 10 points indicating "0": the child is relaxed and calm, "1-3": the child is mildly uncomfortable, "4-6": the child has moderate pain and "7-10": the child has severe pain.
Change from before in anxiety on the CEMS Scale at during peripheral intravenous catheterization | data collected just before and within 5 min after peripheral intravenous catheterization procedure
  The CEMS scale was used to evaluate the anxiety scores of children.This scale, which consists of 5 different categories and 25 items, was used to evaluate the anxiety of children before and during medical procedures. Total score ranges between 5 and 25 points

SECONDARY OUTCOMES:
Change from before in mothers' anxiety on STAI scale at during peripheral intravenous catheterization | data collected just before and within 5 min after peripheral intravenous catheterization procedure
  The STAI scale was used to assess the anxiety mean scores of the mothers.This self-assessment scale with brief statements comprises a total of 40 items, including 20 items in each of two sections, the "state anxiety inventory" and the "trait anxiety inventory". The 'State Anxiety Inventory' was designed to determine what was felt at that moment and the 'Trait Anxiety Scale' was designed to determine what was felt in the last week.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University-Cerrahpaşa, Istanbul
  - Seda Caglar, Istanbul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anderoglu S, Caglar S. The effect of therapeutic play with teddy bear on children's pain, anxiety, and mothers' anxiety during peripheral intravenous catheterisation: a randomised clinical trial. BMC Pediatr. 2025 Dec 6;26(1):29. doi: 10.1186/s12887-025-05769-4. PMID 41351041